CLINICAL TRIAL: NCT00611520
Title: Symbicort in Chronic Obstructive Pulmonary Disease
Acronym: SYMBOL
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Dr Kai Richter, AstraZeneca Germany
Other Study IDs: 1312005009
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: treatment of COPD; related to the budesonide/formoterole therapy in patients with COPD.
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with COPD treated with budesonide/formoterol

SUMMARY:
Under daily routine conditions and without any intervention by the sponsor regarding the selection of subjects, diagnostic procedures, therapeutic decisions (medicinal and non- medicinal therapy, dose, duration, etc.), routine assessments, the participating physicians (i.e. pneumologists and internists) are asked to document relevant data related to the budesonide/formoterole therapy in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD treated with budesonide/formoterol

Exclusion Criteria:

* limitations; possible risks; warnings; contraindications mentioned in the SPC.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 64730 (Actual)
Dates: Start 2005-09; Primary Completion 2005-12 (Actual)

SECONDARY OUTCOMES:
to get further insight into the details of the use , dosage scheme and duration of treatment with budesonide /formoterol in this population

CONTACTS AND LOCATIONS:
Overall Officials: Kai Richter, MD, Study Chair — Medical Department AstraZeneca Germany